CLINICAL TRIAL: NCT00566995
Title: A Phase 2 Study of ZD6474 (Vandetanib) in Patients With Von Hippel Lindau Disease and Renal Tumors
Brief Title: Phase II Study of Vandetanib in Individuals With Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, W. Marston Linehan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080020; 08-C-0020
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Renal Cancer; Von Hippel Lindau
Keywords: Kidney Tumors; Clear Cell Renal Cancer; VEGFR Inhibitor; EGFR Inhibitor; VHL; Von Hippel Lindau; Kidney Tumor
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vandetanib in Participants with Kidney Cancer (Experimental): 300 mg/day (starting dose) oral dose of vandetanib once a day for 28 days
  Interventions: Drug: ZACTIMA (Vandetanib) (ZD6474)

INTERVENTIONS:
Drug: ZACTIMA (Vandetanib) (ZD6474)
  Other Names: Vandetanib

SUMMARY:
This study will examine the effectiveness of an investigational drug called ZD6474 (also known as vandetanib or ZACTIMA). Vandetanib is an experimental drug that is designed to prevent the growth and development of new blood vessels on tumors and to prevent the direct growth of cancer cells. It has been tested in a number of clinical trials on adults with cancer, but the United States (U.S.) Food and Drug Administration has not specifically approved it as a cancer treatment. The purpose of this investigational study is to better understand how vandetanib affects humans who have kidney cancer related to von Hippel-Lindau (VHL) disease, and to develop tests that may improve researchers understanding of kidney cancer and its effects.

Volunteers must be at least 18 years old and must have been diagnosed with kidney cancer related to VHL. Candidates must have a life expectancy greater than three months and must have at least one measurable renal tumor for study purposes. Candidates may not be receiving any other investigational agents or have been treated with an investigational drug within the past four weeks. Candidates who have had surgery, chemotherapy, or radiotherapy within the past four weeks will be excluded from the study. Candidates will be screened with a physical examination and medical history.

During the study, participants will receive an oral dose of vandetanib once a day for 28 days (a treatment period known as a cycle). Participants will need to return to the National Institutes of Health every two weeks on the same day of the week as the first dose of vandetanib for a series of tests and procedures, including blood and urine tests and an electrocardiogram. Every 12 weeks, computerized tomography (CT) or magnetic resonance imaging (MRI) scans will be done to assess the size of participants tumors. Participants whose tumors do not grow and who do not have unacceptable side effects may continue to receive vandetanib to maintain the current condition, until researchers conclude the study....

DETAILED DESCRIPTION:
Background:

Von Hippel Lindau disease is a hereditary cancer syndrome in which affected individuals are at risk for developing tumors in a number of organs, including the kidneys, brain, spine, adrenal glands, eyes and pancreas.

The molecular hallmark of VHL is inactivation of the VHL gene which leads to accumulation of proteins targeted for degradation through the ubiquitin pathway, which includes a group of transcriptionally active proteins called the hypoxia inducible factors (HIF), whose alpha subunits undergo degradation in a VHL-dependent fashion. Accumulation of HIFs results in overexpression of several genes including vascular endothelial growth factor (VEGF), glucose transporter 1 (GLUT-1), transforming growth factor (TGF)-alpha, platelet- derived growth factor (PDGF), and erythropoietin, which are believed to play a role in tumorigenesis, tumor progression and metastasis.

ZD6474 is an orally administered receptor tyrosine kinase inhibitor with activity against the Kinase insert domain-containing receptor/vascular endothelial growth factor receptor 2 (KDR/VEGFR2) and the epidermal growth factor receptor (EGFR). Kinase insert domain receptor (KDR)/vascular growth factor receptor 2 (VEGFR2) is an endothelial cell receptor for vascular endothelial growth factor (VEGF) and plays a crucial role in mediating tumor angiogenesis, while epidermal growth factor receptor (EGFR) (a receptor for TGF-alpha and epidermal growth factor (EGF) is believed to mediate tumor growth and proliferation.

Objective:

Primary Objective

To assess the overall response rate in VHL patients with renal tumors treated with single agent ZD6474

Secondary Objectives:

To study the safety and tolerability of ZD6474

To evaluate time to progression and progression-free survival in VHL patients receiving ZD6474

To study the effect of ZD6474 treatment on non-renal tumors associated with von Hippel Lindau disease ( pancreatic tumors, pheochromocytoma, central nervous system (CNS) hemangioblastomas)

To investigate the effect of ZD6474 on circulating endothelial cells and endothelial progenitor cells and to explore the utility of these markers as surrogates of angiogenesis inhibition

To investigate the effect of ZD6474 on biomarkers of angiogenesis such as plasma VEGF and soluble VEGFR2

Eligibility:

Adults with clinical diagnosis of von Hippel Lindau disease

Presence of one or more measurable renal tumors

Age greater than or equal to 18 years

Adequate organ function, performance status (Eastern Cooperative Oncology Group (ECOG) 0-2) and life expectancy (greater than 3 months)

Design:

Single agent ZD6474 administered daily at a starting dose of 300mg per day

Patients will be evaluated for response every 12 weeks using Response Evaluation Criteria in Solid Tumors (RECIST) criteria

The study is based on an open label two-stage optimal phase II design

Accrual of a maximum of 37 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must satisfy all the following criteria to be eligible for study enrolment.

Clinical diagnosis of von Hippel Lindau disease.

The presence of at least one measurable (as defined by RECIST) renal tumor (renal cell carcinoma (RCC)). Patients with tumors localized to the kidney as well as those with metastatic RCC are eligible.

Age greater than or equal to 18 years.

Life expectancy greater than 3 months

Performance status Eastern Cooperative Oncology Group (ECOG) 0-2.

Patients must have normal organ and marrow function as defined below: white blood cell (WBC) count greater than or equal to 3,000micro/L, absolute neutrophil count greater than or equal to 1,500 micro/L platelet count greater than or equal to 100,000 micro/L, serum creatinine less than or equal to 1.5 times upper limit of reference range or measured 24 hr. creatinine clearance greater than or equal to 50 ml/min, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times upper limit of reference range, total bilirubin less than 1.5 times upper limit of reference range (less than 3 times upper limit of reference range in patients with Gilberts disease), alkaline phosphatase less than or equal to 2.5 times upper limit of reference range (or less than or equal to 5 times upper limit of reference range if considered to be related to liver metastases by the principal investigator (PI)).

No history of serious intercurrent medical illness.

At least four weeks from completion of any other surgical or investigational therapy for von Hippel Lindau and at least 4 weeks from any major surgical procedure. In addition, patients who have undergone recent major surgery should have well healed surgical incisions.

All men and women of childbearing potential must use effective contraception.

Negative pregnancy test in female patients of childbearing potential within 7 days prior to enrolment on study

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Prior or concomitant non-von Hippel Lindau associated malignancy with the exception of adequately treated basal or squamous cell carcinoma of the skin, cervical carcinoma in situ or any other malignancy from which the patient has remained disease free for more than five years.

Known brain metastases (unless adequately resected or irradiated with no evidence of recurrence for at least 6 months).

Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events (to less than or equal to grade 1 Common Terminology Criteria in Adverse Events (CTCAE) v3.0) due to agents administered more than 4 weeks earlier.

Patients may not be receiving any other investigational agents or have received treatment with a non-approved or investigational drug within 4 weeks prior to Day 1 of study treatment except those used for imaging studies.

Use of 5HT-3 antagonists because of the potential effect on corrected QT interval (QTc) interval.

Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes.

Concomitant medications that are potent inducers of cytochrome P450 3A4 (CYP3A4) function, such as rifampin, rifabutin, phenytoin, carbamazepine, barbiturates such as phenobarbital, or St. Johns Wort.

Clinically significant cardiac event (including symptomatic heart failure, myocardial infarction or angina) within 3 months of entry or presence of any cardiac disease that in the opinion of the Principal Investigator increases the risk of ventricular arrhythmia.

History of clinically significant arrhythmia [including multifocal premature ventricular contraction (PVC), bigeminy, trigeminy, ventricular tachycardia] that is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia

Uncontrolled atrial fibrillation. Atrial fibrillation controlled on medication is not excluded.

Presence of Left bundle branch block.

Previous history of QTc prolongation while taking other medications that required discontinuation of that medication.

Congenital long QT syndrome or first degree relative with unexplained sudden death under the age of 40 years QTc with Bazetts correction that is unmeasurable, or greater than or equal to 480 msec on screening electrocardiogram (ECG). If a patient has QTc greater than or equal to 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be less than 480 msec in order for the patient to be eligible for the study). Patients who are receiving a drug that has a risk of QTc prolongation are excluded if QTc is greater than or equal to 460 msec.

Potassium concentration less than 4.0 mEq/L, calcium (ionized calcium or adjusted for albumin), or magnesium concentrations outside normal limits despite optimal supplementation/correction

Left ventricular ejection fraction less than 45 percent measured by multiple gated acquisition scan (MUGA) or echocardiogram (ECHO)

Hypertension not controlled by medical therapy (systolic blood pressure greater than 150 mmHg or diastolic blood pressure greater than 100 mmHg).

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Patient known to be human immunodeficiency virus (HIV) positive and requiring antiretroviral therapy.

Currently active diarrhea that may affect the ability of the patient to absorb ZD6474 or tolerate further diarrhea.

Patients on therapeutic anticoagulation

Patients with known bleeding disorders

Pregnant women are excluded from this study because ZD6474 is an anti-angiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ZD6474, breastfeeding should be discontinued if the mother is treated with ZD6474.

Any known hypersensitivity to ZD6474 or other excipients of ZD6474.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-02-07 (Actual); Primary Completion 2014-06-20 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Marston Linehan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Linehan WM, Lerman MI, Zbar B. Identification of the von Hippel-Lindau (VHL) gene. Its role in renal cancer. JAMA. 1995 Feb 15;273(7):564-70. No abstract available. PMID 7837390
- [Background] Clifford SC, Maher ER. Von Hippel-Lindau disease: clinical and molecular perspectives. Adv Cancer Res. 2001;82:85-105. doi: 10.1016/s0065-230x(01)82003-0. PMID 11447766
- [Background] Kaelin WG Jr. Molecular basis of the VHL hereditary cancer syndrome. Nat Rev Cancer. 2002 Sep;2(9):673-82. doi: 10.1038/nrc885. PMID 12209156
- [Background] Brooks S, Linehan WM, Srinivasan R, Kong HH. Successful laser treatment of vandetanib-associated cutaneous pigmentation. Arch Dermatol. 2011 Mar;147(3):364-5. doi: 10.1001/archdermatol.2011.30. No abstract available. PMID 21422355
- [Background] Vitael, S, Cunningham, D. Meleth, A., Bishop R., Clayton, Datile, M, Linehan WM, Srinivasan R, Meyerle, C. Development of a New Grading System for Corneal Verticillata. ARVO meeting May 8, 2013
- [Background] Vitael, S, Cunningham, D. Meleth, A., Bishop R., Clayton, Datile, M, Linehan WM, Srinivasan R, Meyerle, C. Development of a New Grading System for Corneal Verticillata. ARVO meeting May 2012.
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0020.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vandetanib in Participants With Kidney Cancer
Started | 37
Completed | 30
Not Completed | 7
Not completed — Toxicity | 4
Not completed — Withdrew consent | 3

BASELINE CHARACTERISTICS:
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.65 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate.
Description: Overall response rate is defined as the percentage of participants with either a partial or complete response occurring at any time after initiation of therapy. Response is determined by the Response Evaluation Criteria in Solid Tumors (RECIST). Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Complete response (CR) is a disappearance of all target lesions. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (progressive disease), taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline and every 3 cycles, up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 37
percentage of participants
  Partial Response | 3
  Complete Response | 0
  Stable Disease | 75
  Progressive Disease | 0
  Not Evaluable | 22

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 72 months and 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 37
Participants | 37

3. Secondary Outcome: Time To Progression (TTP)
Description: Time to progression is defined as the time from the start of treatment to progression as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, with death being treated as a censored event. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Complete response (CR) is a disappearance of all target lesions. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, the appearance of one or more new lesions, developing a surgical size tumor that should be resected. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (progressive disease), taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline and every 3 cycles while on study, up to 2 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 37
Months | 13.8 [11.0 to 22.1]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as time from initiation of treatment to either progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria or death. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Complete response (CR) is a disappearance of all target lesions. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (progressive disease), taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline and every 3 cycles while on study, up to 2 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 37
Months | 13.8 [11.0 to 22.1]

5. Secondary Outcome: Effect of Vandetanib (ZD6474) on Endothelial Progenitor Cells
Description: Peripheral blood was collected and analyzed by multiparametric flow cytometry for analysis of angiogenesis markers.
Time Frame: Pre treatment, 4 hours after first treatment, and after one cycle of treatment (one cycle = 28 days)
Population: No samples were received for 2/37 patients.
Measure: Median (Full Range); unit: Cells per 10^6 mononuclear cells
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 35
Cells per 10^6 mononuclear cells
  Cycle 1 Day 1 Pre treatment | 214.44 [0 to 906.7]
  Cycle 1 Day 1, 4 hours post: number analyzed (Participants) | 33
  Cycle 1 Day 1, 4 hours post | 115.79 [0 to 282.69]
  Cycle 2 Day 1: number analyzed (Participants) | 30
  Cycle 2 Day 1 | 160.20 [0 to 640.6]

6. Secondary Outcome: Effect of Vandetanib (ZD6474) on Circulating Endothelial Cells (CEC)
Description: Peripheral blood was collected and analyzed by multiparametric flow cytometry.
Time Frame: Pre treatment, 4 hours after first treatment, and after one cycle of treatment (one cycle = 28 days)
Population: No samples were received for 2/37 participants.
Measure: Median (Full Range); unit: CEC per 10^6 mononuclear cells
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 35
CEC per 10^6 mononuclear cells
  Cycle 1 day 1 Pre treatment | 83.83 [0 to 314.20]
  Cycle 1 Day 1, 4 hours post: number analyzed (Participants) | 33
  Cycle 1 Day 1, 4 hours post | 63.08 [0 to 307.40]
  Cycle 2 Day 1: number analyzed (Participants) | 30
  Cycle 2 Day 1 | 155.8 [0 to 2480]

7. Secondary Outcome: Response in Pancreatic Tumors/Cysts Associated With Von Hippel Lindau (VHL)
Description: Tumor measurements for non-renal tumors were assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) before and after treatment. Tumor measurements for non-renal tumors were assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) before and after treatment. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest um LD recorded since treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline and every 3 cycles while on study, up to 2 years.
Population: Only two participants had target lesions that could be measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 2
Participants
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 0
  Stable Disease | 2

8. Secondary Outcome: Response in Central Nervous System (CNS) Hemangioblastomas Associated With Von Hippel Lindau (VHL)
Description: Tumor measurements for non-renal tumors were assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) before and after treatment. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest um LD recorded since treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline and every 3 cycles while on study, up to 2 years.
Population: Only two participants had target lesions that could be measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 2
Participants
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 0
  Stable Disease | 2

9. Secondary Outcome: Response in Pheochromocytomas Associated With Von Hippel Lindau (VHL)
Description: as for outcome 7
Time Frame: Baseline and every 3 cycles while on study, up to 2 years.
Population: This outcome measure was not done because no participants had measurable lesions.
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Change in Plasma Biomarkers Vascular Endothelial Growth Factor (VEGF) and Soluble Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2) Before and After Treatment With Vandetanib
Description: 5-10cc venous blood was collected for evaluation of basal plasma levels of angiogenesis biomarkers VEGF and VEGFR-2.
Time Frame: Pre treatment, 4 hours after first treatment, and after one cycle of treatment (one cycle = 28 days)
Population: This analysis was intended to be exploratory. Several other studies established that therapy with VEGFR agents modulated serum/plasma VEGF and soluble VEGFR2 levels, but there was no consistent & established correlation with clinical outcome. These analyses were unlikely to add further to our ability to evaluate the major objectives of the study.
Arm/Group | Vandetanib in Participants With Kidney Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 72 months and 14 days
Arm/Group | Vandetanib in Participants With Kidney Cancer
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 5/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib in Participants With Kidney Cancer (N=37)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (3)
Constitutional Symptoms - Other (Specify, generalized weakness) (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Pain - Other (Specify, jaw pain and L shoulder pain) (General disorders) | 1 (1)
Pain::Chest wall (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other, bronchitis; viral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Retinal detachment (Eye disorders) | 1 (2)
Rigors/chills (General disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib in Participants With Kidney Cancer (N=37)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 24 (75)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 17 (37)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 17 (33)
Alkaline phosphatase (Metabolism and nutrition disorders) | 13 (26)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 6 (6)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 5 (8)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 15 (31)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 6 (9)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 (14)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 1 (2) — nonspecific T-wave abnormality
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Constitutional Symptoms - Other (Specify, extreme hunger and jitterness) (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Creatinine (Metabolism and nutrition disorders) | 26 (70)
Cystitis (Renal and urinary disorders) | 2 (2)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (1) — cold sore on lip-herpes simplex
Diarrhea (Gastrointestinal disorders) | 24 (36)
Dizziness (Nervous system disorders) | 5 (7)
Dry eye syndrome (Eye disorders) | 5 (6)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16 (21)
Flatulence (Gastrointestinal disorders) | 3 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 20 (56)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 14 (29)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (4)
Hemoglobin (Blood and lymphatic system disorders) | 5 (10)
Hemoglobinuria (Metabolism and nutrition disorders) | 11 (18)
Hemorrhage, GU::Bladder (Renal and urinary disorders) | 6 (8)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 5 (5)
Hemorrhage, GU::Vagina (Reproductive system and breast disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage/Bleeding - Other (Specify, hematuria) (Renal and urinary disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Cardiac disorders) | 9 (13)
Hypotension (Cardiac disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Infection - Other (Specify, bladder infection) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Dental-tooth (Infections and infestations) | 1 (1)
Insomnia (General disorders) | 11 (16)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (4)
Lymphopenia (Blood and lymphatic system disorders) | 17 (28)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 9 (10)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 16 (37)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Mood alteration::Agitation (Nervous system disorders) | 1 (1)
Mood alteration::Anxiety (Nervous system disorders) | 9 (12)
Mood alteration::Depression (Nervous system disorders) | 6 (6)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Specify, crushed thumb) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (24)
Neurology - Other (Specify, R lower extremity foot weakness) (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (3)
Ocular surface disease (Eye disorders) | 1 (1)
Ocular/Visual - Other (Specify, corneal epithelial defect) (Eye disorders) | 1 (1) — corneal epithelial defect
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1 (1)
Pain - Other (Specify, bilateral ankle pain) (General disorders) | 1 (1) — bilateral ankle pain
Pain::Abdomen NOS (Gastrointestinal disorders) | 2 (4)
Pain::Back (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 3 (4)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain::Oral-gums (Skin and subcutaneous tissue disorders) | 1 (1)
Pain::Pelvis (Reproductive system and breast disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 15 (29)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 4 (9)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 11 (19)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 (7)
Prolonged QTc interval (Cardiac disorders) | 24 (119)
Proteinuria (Metabolism and nutrition disorders) | 21 (44)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (3)
Pulmonary/Upper Respiratory - Other (Specify, asthma) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (7)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 30 (48)
Renal/Genitourinary - Other (Specify, hematuria) (Renal and urinary disorders) | 1 (1)
Seroma (Musculoskeletal and connective tissue disorders) | 1 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 14 (25)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 1 (2)
Sweating (diaphoresis) (General disorders) | 3 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 (2)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 13 (32)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (4)
Vision-blurred vision (Eye disorders) | 2 (2)
Vision-flashing lights/floaters (Eye disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (8)
Weight gain (General disorders) | 2 (3)
Weight loss (General disorders) | 9 (14)
Cardiac arrhythmia-Other, Specify (tachycardia) (Cardiac disorders) | 1 (1)
Dermatology/Skin - Other (Specify, dry scalp) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify,dry, chapped lips) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify,eczematous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify, erythema L leg) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify, erythema on face) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify, paronychia of L great toe) (Skin and subcutaneous tissue disorders) | 1 (1)
Infection - Other (Specify, bladder (urinary) (Infections and infestations) | 1 (1)
Infection - Other (Specify, sinusitis) (Infections and infestations) | 1 (1)
Infection - Other (Specify, tooth abscess) (Infections and infestations) | 1 (1)
Infection - Other (Specify, sinus infection) (Infections and infestations) | 1 (1)
Ocular/Visual - Other (Specify, corneal verticillata) (Eye disorders) | 1 (1)
Ocular/Visual - Other (Specify, halos at night) (Eye disorders) | 1 (1)
Ocular/Visual - Other (Specify, ocular/visual other-vortex keratopathy) (Eye disorders) | 1 (1)
Pain - Other (Specify, cramp in extremities) (General disorders) | 1 (1)
Pain - Other (Specify, dysuria) (General disorders) | 1 (1)
Pain - Other (Specify, intermittent chest/thorax) (General disorders) | 1 (1)
Pain - Other (Specify, left elbow) (General disorders) | 1 (1)
Pain - Other (Specify, myalgia) (General disorders) | 1 (1)
Pain - Other (Specify, pain bilateral feet) (General disorders) | 1 (1)
Pain - Other (Specify, pain under R ribcage) (General disorders) | 1 (1)
Pain - Other (Specify, pain-L elbow pain) (General disorders) | 1 (1)
Pain - Other (Specify, pain-R ankle pain) (General disorders) | 1 (1)
Pain - Other (Specify, R shoulder) (General disorders) | 1 (1)
Pain - Other (Specify, suprapubic) (General disorders) | 1 (1)
Pain - Other (Specify, tooth sensitivity) (General disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, bronchitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, cold) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, cold symptoms) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, congestion) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, upper respiratory infection) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/Genitourinary - Other (Specify, LUTS Syndrome - decreased urinary flow) (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Other (Specify, microscopic hematuria) (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2012-03-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT00566995/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT00566995/Prot_SAP_001.pdf